CLINICAL TRIAL: NCT05253625
Title: The Effect of Lullaby Listened to Preterm Babies in Neonatal Intensive Care Units on Physiological Parameters and Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Izmir Tinaztepe University (Other)
Responsible Party: Principal Investigator, Nilüfer Özgürbüz, Ass. Prof.Dr. Nilüfer Özgürbüz, Izmir Tinaztepe University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: IzmirTinaztepeU NOzgurbuz
Record Dates: First submitted 2022-01-31; First posted 2022-02-24 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Neonatal Intensive Care; Music Therapy; Pain Responses
Keywords: premature; pain; lullaby
MeSH Terms: conditions — Premature Birth; Pain

STUDY DESIGN:
Intervention Model Description: The participants will be assigned to three groups. Before, during and after a painful intervention the first group (Group A) will listen to a lullaby recorded with the mothers voice, the second group (Group B) will listen to a lullaby recorded with a unfamiliar female voice, and the third group (Group C) without and intervention (no lullaby).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- lullaby mother (Experimental): The participant will listen to a lullaby recorded with his mothers voice.
  Interventions: Other: Listening to a recorded lullaby.
- lullaby female (Experimental): The participant will listen to a lullaby recorded with a foreign female voice.
  Interventions: Other: Listening to a recorded lullaby.
- no lullaby (No Intervention): The participant will not listen to a lullaby.

INTERVENTIONS:
Other: Listening to a recorded lullaby. — A lullaby will be played from the MP4 player on the outer foot of an empty incubator, and a decibel meter (dB) will be placed in the empty incubator, so that the maximum level of the decibel meter does not exceed 50-60 dB (45-65 dB according to APA). ) (American Academy of Pediatrics. ACOG.2007) (Guidelines for Pediatrics Care. 7th edition) sound adjustment will be made. The lullaby with the mother's voice (first arm newborn mothers) adn with an unfamiliar female voice (second arm newborns) will be recorded in MP4 beforehand. The lullabies of groups A and B are lullabies performed in approximately 4 minutes and will be played repeatedly for the specified periods.
  Arms: lullaby female; lullaby mother

SUMMARY:
Preterms who enter a different environment after the intrauterine period experience an adaptation process and may need special care due to conditions such as developmental disabilities or neurological disorders. In such cases, newborns may frequently be exposed to repetitive painful interventions (like IV catherization). Pain in the postnatal period can cause physiological, behavioral and metabolic changes, and changes in the functional processing related with somatosensation and pain in the long term. In this context, inadequacy in pain control may cause neurodevelopmental and behavioral problems in infants.

For these reasons, it is essential to carefully evaluate the pain status of the newborn and to perform pharmacological and/or non-pharmacological interventions. In the intrauterine 20th week, the ability to hear begins to form, and in the 26-28th weeks the level to respond to sounds is achieved. Music therapy is a method that can be used for newborns as it reaches a level that can respond to sound stimuli within weeks. Especially in the 32nd gestational week, preterm newborns begin to develop the ability to distinguish mother's voice from other sounds with regard to rhythm and intonation. Due to this developmental feature of preterm newborns, it is recommended to use the mother's voice in neonatal intensive care units. However, studies on this subject are very limited.

The main goal of care in neonatal intensive care units is to maintain the baby's life and comfort at the highest level, to minimize pain and suffering, and to ensure that it can cope with pain. In the light of all information, it is essential to strengthen scientific evidence in order to apply non-pharmacological methods in clinics. The research was planned experimentally in order to examine the effects of listening to a lullaby on pain and physiological parameters in preterms hospitalized in neonatal intensive care units. The participants will be devided in three groups. The first group will listen to the lulliby recorded with the mothers voice, the second group will listen to the the lulliby recorded with the voice of an unfamilliar female, and the third group will not listen to a lulliby. The effects will be measured by using three physiologic parameters (oxygen saturation, heart rate, and respiratory rate) and pain responses (Neonatai Infant Pain Scala) before, during, and after a painful intervention (IV catherization).

ELIGIBILITY:
Inclusion Criteria:

* At 32-36+6 weeks of gestation
* Stable first 24 hours after birth
* Not dependent on mechanical ventilation
* Non-intubated
* Without a congenital and/or acquired malformation of hearing
* No congenital defect • Without hyperbilirinemia
* Not taking analgesics and/or sedatives in the last 24 hours
* If no painful application has been made to the newborn in the last hour (eg, blood collection, aspiration, eye examination, etc.)
* Postnatal age of 1-7 days
* Preterms whose height and weight are above the 10% percentile according to the week of gestation

Exclusion Criteria:

* Deterioration in general condition
* Those who do not meet the criteria for inclusion in the research
* Preterms whose parents did not consent to participate in the study

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Estimated)
Dates: Start 2022-03-08 (Estimated); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of NIPS (Neonatal Infant Pain Scale) Score | 15 minutes before the IV cateherization, 2 minutes before the catherization, during the catherization, 3 minutes after the catherization, and 15 minutes after the catherization.
  Pain response according to Neonatal Infant Pain Scale
Change of SpO2 (Oxygen Concentration) | 15 minutes before the IV cateherization, 2 minutes before the catherization, during the catherization, 3 minutes after the catherization, and 15 minutes after the catherization.
  Oxygen saturation
Change of HR (Heart Rate) | 15 minutes before the IV cateherization, 2 minutes before the catherization, during the catherization, 3 minutes after the catherization, and 15 minutes after the catherization.
  Heart rate
Change of RR (Respiratory Rate) | 15 minutes before the IV cateherization, 2 minutes before the catherization, during the catherization, 3 minutes after the catherization, and 15 minutes after the catherization.
  Respiratory rate

CONTACTS AND LOCATIONS:
Overall Officials: Nilüfer Özgürbüz, PhD, Principal Investigator — Izmir Tinaztepe University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cignacco E, Hamers JP, Stoffel L, van Lingen RA, Gessler P, McDougall J, Nelle M. The efficacy of non-pharmacological interventions in the management of procedural pain in preterm and term neonates. A systematic literature review. Eur J Pain. 2007 Feb;11(2):139-52. doi: 10.1016/j.ejpain.2006.02.010. Epub 2006 Apr 3. PMID 16580851
- [Background] de Melo GM, Lelis AL, de Moura AF, Cardoso MV, da Silva VM. [Pain assessment scales in newborns: integrative review]. Rev Paul Pediatr. 2014 Dec;32(4):395-402. doi: 10.1016/j.rpped.2014.04.007. PMID 25511005
- [Background] Halimaa SL, Vehvilainen-Julkunen K, Heinonen K. Knowledge, assessment and management of pain related to nursing procedures used with premature babies: questionnaire study for caregivers. Int J Nurs Pract. 2001 Dec;7(6):422-30. doi: 10.1046/j.1440-172x.2001.00322.x. PMID 11785445
- [Background] Yigit S, Ecevit A, Koroglu OA. Turkish Neonatal Society guideline on the neonatal pain and its management. Turk Pediatri Ars. 2018 Dec 25;53(Suppl 1):S161-S171. doi: 10.5152/TurkPediatriArs.2018.01802. eCollection 2018. PMID 31236029
- [Background] American Academy of Pediatrics Committee on Fetus and Newborn; American Academy of Pediatrics Section on Surgery; Canadian Paediatric Society Fetus and Newborn Committee; Batton DG, Barrington KJ, Wallman C. Prevention and management of pain in the neonate: an update. Pediatrics. 2006 Nov;118(5):2231-41. doi: 10.1542/peds.2006-2277. PMID 17079598
- [Background] Levitin DJ, Tirovolas AK. Current advances in the cognitive neuroscience of music. Ann N Y Acad Sci. 2009 Mar;1156:211-31. doi: 10.1111/j.1749-6632.2009.04417.x. PMID 19338510
- [Background] Bieleninik L, Ghetti C, Gold C. Music Therapy for Preterm Infants and Their Parents: A Meta-analysis. Pediatrics. 2016 Sep;138(3):e20160971. doi: 10.1542/peds.2016-0971. Epub 2016 Aug 25. PMID 27561729
- [Background] Dehaene-Lambertz G, Montavont A, Jobert A, Allirol L, Dubois J, Hertz-Pannier L, Dehaene S. Language or music, mother or Mozart? Structural and environmental influences on infants' language networks. Brain Lang. 2010 Aug;114(2):53-65. doi: 10.1016/j.bandl.2009.09.003. Epub 2009 Oct 27. PMID 19864015
- [Background] Standley JM. A meta-analysis of the efficacy of music therapy for premature infants. J Pediatr Nurs. 2002 Apr;17(2):107-13. doi: 10.1053/jpdn.2002.124128. PMID 12029604
- [Background] Cevasco AM. The effects of mothers' singing on full-term and preterm infants and maternal emotional responses. J Music Ther. 2008 Fall;45(3):273-306. doi: 10.1093/jmt/45.3.273. PMID 18959452
- [Background] Loewy J, Stewart K, Dassler AM, Telsey A, Homel P. The effects of music therapy on vital signs, feeding, and sleep in premature infants. Pediatrics. 2013 May;131(5):902-18. doi: 10.1542/peds.2012-1367. Epub 2013 Apr 15. PMID 23589814
- [Background] Vianna MN, Barbosa AP, Carvalhaes AS, Cunha AJ. Music therapy may increase breastfeeding rates among mothers of premature newborns: a randomized controlled trial. J Pediatr (Rio J). 2011 May-Jun 8;87(3):206-12. doi: 10.2223/JPED.2086. Epub 2011 Apr 1. English, Portuguese. PMID 21461451